CLINICAL TRIAL: NCT05854667
Title: Addition of High Dose Stimulant and Engagement-focused Contingency Management (CM), Alone and in Combination, to Treatment as Usual (TAU) for the Management of Methamphetamine (MA) Use Disorder (ASCME): a Canadian Multi-centre, RCT
Brief Title: Clinical Trial of High Dose Lisdexamfetamine and Contingency Management in MA Users
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 23.053
Record Dates: First submitted 2023-04-06; First posted 2023-05-11 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12

CONDITIONS: Methamphetamine Abuse; Methamphetamine-dependence; Addiction, Substance; Addiction
Keywords: Contingency Management; Treatment as Usual
MeSH Terms: conditions — Substance-Related Disorders; Behavior, Addictive | interventions — Therapeutics; Lisdexamfetamine Dimesylate

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of four arms:
  1. Treatment as Usual with Placebo
  2. Treatment as Usual with Placebo and Contingency Management
  3. Treatment as Usual with Lisdexamfetamine (LDX-01)
  4. Treatment as usual with Lisdexamfetamine (LDX-01) and Contingency Management
Who Masked: Participant, Care Provider, Investigator
Masking Description: All participants will receive identical capsules (i.e., smell, taste, and colour), reducing bias by blinding participants, providers, and research staff to the study drug.
  To maintain the blinding of the study medication, dose adjustments will be known by Qualified Investigators and the Pharmacy team according to the Induction Phase schedule and at the Investigator's discretion, without unblinding the study medication (i.e., LDX-01 versus placebo) except for some limited safety related reasons. Access to the randomization code will be strictly controlled by the Data Management Centre. Each participant's assignment will be kept so that an individual code may be broken without unblinding the randomization allocation of other participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Treatment as Usual plus Placebo (Placebo Comparator): Participants will receive treatment as usual at the clinic as well as once daily lisdexamfetamine matched Placebo orally for 15 weeks.
  Interventions: Drug: Treatment as Usual plus Placebo
- Treatment as Usual plus Placebo plus Contingency Management (Placebo Comparator): Participants will receive treatment as usual at the clinic, once daily lisdexamfetamine matched placebo medication orally for 15 weeks, as well as engagement-focused contingency management.
  Interventions: Drug: Treatment as Usual plus Placebo plus Contingency Management
- Treatment as Usual plus lisdexamfetamine (LDX-01) (Active Comparator): Participants will receive treatment as usual at the clinic as well as once daily over-encapsulated lisdexamfetamine (LDX-01) orally for 15 weeks.
  Interventions: Drug: Treatment as Usual plus lisdexamfetamine (LDX-01)
- Treatment as Usual plus lisdexamfetamine (LDX-01) plus Contingency Management (Active Comparator): Participants will receive treatment as usual at the clinic, once daily over-encapsulated lisdexamfetamine (LDX-01) orally for 15 weeks, as well as engagement-focused contingency management.
  Interventions: Drug: Treatment as Usual plus lisdexamfetamine (LDX-01) plus Contingency Management

INTERVENTIONS:
Drug: Treatment as Usual plus Placebo — Participants receive once daily Lisdexamfetamine matched placebo for 15 weeks, as well as treatment as usual at clinical site.
  Other Names: Contingency Management
  Arms: Treatment as Usual plus Placebo
Drug: Treatment as Usual plus Placebo plus Contingency Management — Participants receive once daily Lisdexamfetamine matched placebo for 15 weeks, as well as treatment as usual at clinical site, and engagement-focused contingency management for 12 weeks, week 2-13.
  Arms: Treatment as Usual plus Placebo plus Contingency Management
Drug: Treatment as Usual plus lisdexamfetamine (LDX-01) — Participants receive once daily Lisdexamfetamine for 15 weeks, as well as treatment as usual at clinical site. Medication is provided in 3 phases:
  Week 1 (Induction Phase): 100 mg (Day 1 and 2), 150 mg (Day 3 and 4), 200 mg (Day 5, 6 and 7) Weeks 2-13 (Maintenance Phase): 250 mg per day (or the maximum tolerated for each individual) and then will continue on the same daily dose Weeks 14-15 (Taper Phase): 150 mg (Week 14) and 50 mg (Week 15).
  Arms: Treatment as Usual plus lisdexamfetamine (LDX-01)
Drug: Treatment as Usual plus lisdexamfetamine (LDX-01) plus Contingency Management — Participants receive once daily Lisdexamfetamine for 15 weeks, as well as treatment as usual at clinical site. Medication is provided in 3 phases:
  Week 1 (Induction Phase): 100 mg (Day 1 and 2), 150 mg (Day 3 and 4), 200 mg (Day 5, 6 and 7) Weeks 2-13 (Maintenance Phase): 250 mg per day (or the maximum tolerated for each individual) and then will continue on the same daily dose Weeks 14-15 (Taper Phase): 150 mg (Week 14) and 50 mg (Week 15). Engagement-focused contingency management will be provided for 12 weeks, Week 2-13.
  Other Names: Contingency Management
  Arms: Treatment as Usual plus lisdexamfetamine (LDX-01) plus Contingency Management

SUMMARY:
The goal of this clinical trial is to learn if administering a high dose stimulant with Contingency Management reduces days of use in adults who use methamphetamine better than the usual treatment provided by the clinic.

The main questions the trial aims to answer are:

Is a high dose stimulant better than a placebo and usual treatment at helping reduce the number of days they use methamphetamine? Is a high dose stimulant with contingency management better than placebo and usual treatment at helping people reduce the number of days they use methamphetamine?

Participants will be placed randomly into one of four groups:

1. Usual treatment and placebo
2. Usual treatment, placebo and contingency management
3. Usual treatment and high dose stimulant
4. Usual treatment, high dose stimulant and contingency management

Participation includes the following:

1. Participants will receive medication or placebo weekly for 15 weeks.
2. Participants will attend the clinic for weekly treatment
3. Participants will attend the clinic once every 2 weeks for study visits. Each visit will take about an hour to complete. At these visits, participants will be asked to provide a urine sample and complete questionnaires.

DETAILED DESCRIPTION:
The ASCME trial is a multi-centre, randomized double blind (lisdexamfetamine-01 component), open label (Contingency Management component), dose-ascending, placebo controlled trial. Participants will be enrolled in one of the 4 treatment arms:

Arm 1: treatment as usual plus placebo Arm 2: treatment as usual plus placebo and contingency management Arm 3: treatment as usual plus lisdexamfetamine (LDX-01) Arm 4: treatment as usual plus lisdexamfetamine (LDX-01) and contingency management

The trial will enroll 440 participants, and will be conducted in 5-7 treatment centres across Canada.

Participants will be enrolled in the trial for 20 weeks altogether.

ELIGIBILITY:
Inclusion Criteria:

* Participant must meet all the following criteria:

  1. Between 18 and 55 years of age;
  2. Diagnosed with a moderate to severe methamphetamine (MA) use disorder as defined by the DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, 5th edition) criteria;
  3. Active MA use at screening measured via self-reported MA use ≥14 days in the past 28 days AND verified by urine drug metabolite testing;
  4. Interested in reducing/stopping MA use;
  5. If female:

     1. Be of non-childbearing potential, defined as (i) postmenopausal (12 months of spontaneous amenorrhea and ≥ 45 years of age); or (ii) documented surgically sterilized (i.e., tubal ligation, hysterectomy, or bilateral oophorectomy); or
     2. Be of childbearing potential, have a negative pregnancy test at screening, and agree to use an acceptable method of birth control throughout the study;
  6. Willing to be randomized to one of the 4 study arms and followed for the duration of the trial;
  7. Able to provide informed consent;
  8. Willing to comply with study procedures;
  9. Able to communicate in English or French.

Exclusion Criteria:

* 1. Symptomatic or advanced cardiovascular disease (e.g., advanced arteriosclerosis), moderate hypertension; current hyperthyroidism confirmed via blood test; known hypersensitivity or idiosyncrasy to the sympathomimetic amines or glaucoma or any disabling, severe, OR unstable medical condition that, in the opinion of the study physician, precludes safe participation or the ability to provide fully informed consent; 2. Any severe or unstable co-morbid substance use disorder that, in the opinion of the study physician, precludes safe participation in the study; 3. Participants with Opioid Use Disorder (OUD) who have been on Opioid Agonist Therapy (OAT) for < 12 weeks, and not yet at stabilization dose, or at stabilization dose < 4 weeks; 4. Current or history of any serious psychiatric disorder (e.g., bipolar disorder, pre-existing psychosis, schizophrenia) that, in the opinion of the study physician, precludes safe participation in the study; 5. History of a severe adverse event, hypersensitivity or known allergic reaction to LDX or other amphetamine drugs OR hypersensitivity to the sympathomimetic amines; 6. Pregnant, nursing, or planning to become pregnant during the study period; 7. Planned extended absence during study period (e.g., pending legal action, surgery, incarceration, inpatient residential program) in the opinion of the study physician that might prevent completion of the study; 8. Use of an investigational drug for stimulant use disorder during the 30 days prior to screening, confirmed via self-report OR pharmacy records; 9. Currently receiving contingency management for the treatment of stimulant use disorder in the 4 weeks prior to screening, confirmed via self-report OR site records; 10. Use of prescribed amphetamine-type medication OR medication for the treatment of stimulant use disorder (e.g., methylphenidate, modafinil, bupropion) in the 4 weeks prior to screening; 11. Current or anticipated need for treatment with any medication that may interact with LDX (e.g., proton pump inhibitors, monoamine oxidase inhibitors [MAOIs]) used currently or within the past 14 days AND that would preclude study participant at the discretion of the study physician

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 440 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Total number of days of methamphetamine use during maintenance phase | 12 weeks
  The primary outcome measure is the total number of days of MA use during the 12-week maintenance treatment period of the trial, assessed via self-report using the Timeline Followback (TLFB) Questionnaire.

SECONDARY OUTCOMES:
Medication Adherence | 15 weeks
  Medication adherence will be measured by the number of days the medication is taken as prescribed. The medication is provided to the patient in Blister Packaging, with an electronic data monitoring system affixed. The date and time each dose is taken by participant will be recorded by the electronic blister pack database. This data will be extracted from an Electronic Blister Packaging Database, and pharmacy abstraction. Retention on study medication/placebo will be defined as the proportion of participants (LDX-01 or placebo) at D1 of Week 15, having an active prescription for the treatment, confirmation via self-report by the participant of ingestion of medication/placebo and monitoring of the electronic blister pack.
Safety Events | 20 weeks
  Safety in the trial will be evaluated by monitoring adverse events and serious adverse events over the entire course of the study; (i.e., baseline (Day 1), Day 3, and Day 5 of Week 1, and Day 1 of Weeks 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 16, and 20 (end of follow-up). Adverse events and serious adverse events will be defined and documented according to the adverse reporting procedures.Information regarding safety events will be collected via self-report, report from others, or chart abstraction, or all of the above.
Changes in Quality of Life | Will be administered at Baseline, Week 8, 14 and 20.
  Quality of life will be measured using the WHO Quality of Life-BREF40 which is person-centred generic patient-reported quality of life measure, being validated to document and follow changes in quality of life in different physical and psychiatric disorders. It specifically looks at 4 domains related to quality of life: physical health, psychological health, social relationships, and environment. Quality of Life Assessment will yield data on the number of participants that report more positive quality of life in the domains of physical health, psychological health, social relationships, and environment.
Methamphetamine and other Substance Use - self report | 15 weeks
  Methamphetamine and other substance use will be measured every two weeks by self report using the time line follow back (TLFB). The TLFB collects self-reported substance use amount, frequency, and duration retrospectively over the past 14 days. The TLFB has shown very good reported psychometric properties in adults using substances.
Methamphetamine and other Substance Use - urine drug screen | 15 weeks
  Urine samples for drug screens will be collected at screening, baseline, and every 2 weeks for the 12- week Maintenance Phase, as well during the taper and follow-up phases. All urine specimens will be collected and analysed using Health Canada approved, Rapid Response Multi-Drug One Step Screen Test Panel, and will follow all manufacturer's recommended procedures to test for the presence of the following drugs or their respective metabolites: amphetamine, methamphetamine, morphine, fentanyl, benzodiazepines, cocaine, THC, methadone, buprenorphine, methylphenidate, MDMA, LSD, ketamine, oxycodone, heroin, Hydromorphone. A further validity check will be performed using a commercially available adulterant test strip.
Indigenous wellness perspective | Administered at Baseline, week 8, 14 and 20
  The Wellness Registry Tool - 10 (WRT-10) aims to capture the voice of Indigenous participants with respect to their own wellness, in a culturally relevant way, with the broader goal to improve mental, physical, emotional, and spiritual wellness. This tool has 3 sections: 1) aspects of balance: physical, mental emotional and spiritual health and well-being, 2) Social connectedness, and 3) participation in cultural practices. Section 1 & 2 are rated on a 5-point Likert scale and captures how participants rate their overall (holistic) wellbeing, as well as each individual component of their wellbeing. Section 3 captures participant engagement with cultural activities, services, supports, and healing traditions.
Treatment Satisfaction | Week 14 only
  Treatment satisfaction will be assessed using the Client Satisfaction Questionnaire-8 (CSQ-8) and has shown good psychometric properties (Matsubara et al., 2013). The CSQ-8 collects information on the participant's satisfaction as it relates to the assigned medication and the clinical care received at the site.

CONTACTS AND LOCATIONS:
Overall Officials: Didier Jutras-Aswad, Principal Investigator — University of Montreal Hospital Research Center
Locations (4):
- Canada (4):
  - Rapid Access Addiction Medicine Clinic, St. Paul's Hospital, Vancouver, British Columbia
  - River Stone Recovery Centre, Fredericton, New Brunswick
  - Center for Addiction and Mental Health, Toronto, Ontario
  - University of Montreal Hospital Research Center, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No